CLINICAL TRIAL: NCT02586272
Title: A Prospective, Single-center, Randomized, Two-arm, Interventional Study to Evaluate the Implantation Rate of Embryos Selected on the Basis of Morphology and Granulocyte-Colony Stimulating Factor (G-CSF) Concentration in the Ovarian Follicular Fluid (FF) - FF G-CSF - Compared to the Implantation Rate of Embryos Selected on the Basis of Morphology Alone When Elective Single Embryo Transfer (SET) of a Fresh Embryo is Performed on Day 2/3 After Oocyte Retrieval.
Brief Title: Diafert for Embryo Selection and Fertility Improvement
Acronym: DESTINy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0040-100; 2014-001635-36 (EudraCT Number)
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Infertility
Keywords: Embryo Transfer; assisted reproductive technology
MeSH Terms: conditions — Infertility | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daifert (Experimental): • Interventional Group: The embryo to be transferred is selected on the basis of both morphological assessment performed on Day 2 or 3 and FF G-CSF concentration. FF G-CSF concentration will be measured with the Diafert® immunoassay.
  Interventions: Device: Daifert
- Control Group (Other): Control Group: The embryo to be transferred is selected on the basis of morphological assessment performed on Day 2 or 3.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Device: Daifert
  Arms: Daifert
Procedure: Control Group
  Other Names: Control - Morphological Assessment
  Arms: Control Group

SUMMARY:
Prospective, single-center, single-blind, randomized, controlled, two-arm, interventional study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women at least 18 years old at the time of informed consent.
* 2. Able to understand and voluntarily sign an Informed Consent form approved by the relevant Independent Ethics Committee (IEC) governing the site.
* 3. First or second fresh Assisted Reproductive Technology (ART) cycle attempt (since last successful implantation, if any).
* 4. Eligible for elective SET of fresh embryo on Day 2/3. Elective SET is defined as a transfer for which there is more than one embryo in the same morphological ("best") category as that of the selected embryo.

Exclusion Criteria:

* 1. Presence or history of ovarian endometriotic cyst.
* 2. Presence or history of diagnosed severe endometriosis (i.e. stage IV the revised American Fertility Society classification for endometriosis).
* 3. Hormonal, functional, anatomical and/or any other abnormalities potentially increasing the risk of miscarriage and/or ectopic pregnancy as judged by the Investigator and determined by medical history and clinical laboratory. This includes, but is not limited to, uncontrolled diabetes mellitus, uncontrolled thyroid disease, alcoholism, drug abuse, abnormal uterine cavity etc.
* 4. History of two or more consecutive miscarriages.
* 5. Known history of human immunodeficiency virus, Hepatitis C virus and/or Hepatitis B virus infection.
* 6. The subject has other serious or acute conditions that, in the Investigator's opinion, would preclude her participation in the study.
* 7. Need for preimplantation genetic diagnosis/screening.
* 8. Use of time-lapse embryo imaging.
* 9. Participating in oocyte donation procedure.
* 10. Participation in any interventional drug clinical investigation within 2 months prior to screening.
* 11. Dependency on sponsor or investigator (e.g. co-worker or family member).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Percentage of successful implantations | At Week 6
  The percentage of successful implantation 6 weeks after oocyte retrieval (±3 days), i.e. at approximately 8 weeks gestational age (±3 days) or 8 weeks of amenorrhea (± 3 days), in each group (Control and Interventional groups), overall and within each morphological embryo category, when elective Single Embryo Transfer (SET) is performed on Day 2 or 3.
  Successful implantation is defined as the presence in the uterus of at least one gestational sac with fetal heart activity identified on ultrasound.

SECONDARY OUTCOMES:
Percentage of live births | Approximately Week 40 (pregnancy outcome)
  Percentage of live birth in the Control group and in the Interventional group when elective SET of a fresh embryo is performed on Day 2 or 3 after oocyte retrieval.

CONTACTS AND LOCATIONS:
Overall Officials: Tennador Sanderson, Study Director — Forest Laboratories, an affiliate of Allergan plc
Locations (1):
- Leuven University Fertility Center, Leuven, Belgium